CLINICAL TRIAL: NCT04411862
Title: Efficacy of Phosphatidylcholine in Addition to Behavior Therapy by Clinical Pharmacist in the Management of Non Alcoholic Fatty Liver (NAFLD)
Brief Title: Efficacy of Phosphatidylcholine in NAFLD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nehal Abou Seada (Other)
Responsible Party: Sponsor-Investigator, Nehal Abou Seada, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD
Record Dates: First submitted 2020-05-10; First posted 2020-06-02 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Phosphatidylcholines; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Shams University Hospitals and Ain Shams Specialized Hospital outpatient Gastroenterology Clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 50 Participants with NAFLD that receive lifestyle modification by Clinical Pharmacist plus Phosphatidylcholine two soft capsules 3 times daily(2.1 g per day) for 6 month
  Interventions: Dietary Supplement: Phosphatidyl Choline; Behavioral: Lifestyle modification
- Control Group (Active Comparator): 50 Participants with NAFLD that receive only lifestyle modification by Clinical Pharmacist
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Dietary Supplement: Phosphatidyl Choline — 2.1 g Phosphatidylcholine daily in addition to lifestyle modification
  Arms: Intervention Group
Behavioral: Lifestyle modification — Lifestyle modification and health education by Clinical Pharmacist
  Other Names: Behavior therapy; Health education

SUMMARY:
This study evaluates efficacy of Phosphatidylcholine in addition to life style modification and patient health education by clinical Pharmacist in the Management of Non Alcoholic Fatty Liver NAFLD. All participants with NAFLD will receive life style intervention and half of them will receive additionally Phosphatidylcholine.

DETAILED DESCRIPTION:
As a result of increasing rates of obesity Non Alcoholic Fatty Liver (NAFLD) is the most common liver disorder affecting 17-46% of adults and parallels the prevalence of Metabolic Syndrome (MetS) and its components which also increases the risk of more advanced disease both in adults and in children.

Its pathogenesis is complex and multifactorial, mainly involving genetic, environmental and metabolic factors. New concepts are constantly appearing in the literature, promising new diagnostic and therapeutic tools. Further studies are needed to better characterize not only NAFLD development but overall NAFLD progression, in order to better identify NAFLD patients at higher risk of metabolic, cardiovascular and neoplastic complications. Pharmacological treatments aimed primarily at improving liver disease should generally be limited to those with biopsy-proven Nonalcoholic steatohepatitis (NASH) and liver ﬁbrosis. Not much therapeutic options for NAFLD are accepted until today besides correction of obesity with hypocaloric diets and physical exercise and controlling hyperglycemia with diet, insulin, or oral hypoglycemic agents. Weight loss generally reduces hepatic steatosis.Essential phospholipid (EPL) as a nutritional supplement is one of the drugs under discussion with significant positive effects as antioxidative, antifibrotic effects and high biocompatibility on NAFLD.

ELIGIBILITY:
Patients were included in the study when the following criteria to were fulfilled :

Inclusion Criteria:

* fatty liver upon Ultrasonography (US) /Computed Tomography (CT) /Magnetic Resonance Imaging (MRI) with either incidental increased Alanine Aminotransferase (ALT)
* the presence of risk factors related to NAFLD + increased ALT
* symptomatic liver disease +/- hepatomegaly, +/- increased ALT
* homeostasis model assessment-insulin resistance HOMA IR score > 3
* presence of liver steatosis or stiffness measured by transient elastography
* eligible patients had at least one of the following metabolic comorbidities: hypertension, Type 2 Diabetes Mellitus, overweight/obesity (BMI>27 kg/m2) serum cholesterol of > 200 mg/d

Patients were excluded from the study if showing evidence :

Exclusion Criteria:

* if showing evidence of alcoholic or chronic liver disease
* Hepatocellular Carcinoma, autoimmune hepatitis
* end stage liver disease
* treatment with other hepatoprotectants
* other concomitant EPL within 30 days of study initiation
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
change from baseline Body Mass Index (BMI) at 3 and 6 month | baseline, at 3 and 6 month
  person's weight in kilograms divided by the square of the person's height in metres (kg/m2).
change from baseline liver stiffness at 3 and 6 month | baseline , at 3 and 6 month
  Liver Stiffness and fibrosis score measured by Transient elastography (Fibroscan) F0 = no fibrosis F1 = portal fibrosis without septa F2 = portal fibrosis with few septa F3 = numerous septa without cirrhosis F4 = cirrhosis
change from baseline Lipid Profile | baseline , at 3 and 6 month
  Total cholesterol ,Triglyceride ,Low Density Lipoprotein ,High Density Lipoprotein
change from baseline Oxidative stress markers | baseline , at 3 and 6 month
  malonaldehyde (MDA) as an index of lipid peroxidation by colorimetric assay
change from baseline NAFLD score at 3 and 6 month | baseline , at 3 and 6 month
  NAFLD Fibrosis Score is based on six readily available variables (age, BMI, hyperglycemia, albumin, platelet count, AST/ALT ratio) and it is calculated using published formula (http: //naflds- core.com) . A low cutpoint (score < -1.455) signified the absence of advanced fibrosis, whereas a high cutpoint (score> 0.676) identified advanced fibrosis.
change from baseline homeostasis model assessment Insulin resistance HOMA IR scores at 3 and 6 month | baseline , at 3 and 6 month
  HOMA IR scores <3 normal HOMA IR scores >5 severe insulin resistance 3 to 5 moderate insulin resistance

SECONDARY OUTCOMES:
change from baseline Complete Blood Picture at 3 and 6 month | baseline , at 3 and 6 month
  platelet count

REFERENCES:
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Chalasani N; Writing Group for American Association for Study of Liver Diseases; American College of Gastroenterology; American Gastroenterology Association practice guideline on Diagnosis and Management of Nonalcoholic Fatty Liver Disease. Reply: To PMID 22488764. Hepatology. 2013 Feb;57(2):853-4. doi: 10.1002/hep.26199. Epub 2013 Jan 7. No abstract available. PMID 23297154
- [Background] Ahmed MH, Noor SK, Bushara SO, Husain NE, Elmadhoun WM, Ginawi IA, Osman MM, Mahmoud AO, Almobarak AO. Non-Alcoholic Fatty Liver Disease in Africa and Middle East: An Attempt to Predict the Present and Future Implications on the Healthcare System. Gastroenterology Res. 2017 Oct;10(5):271-279. doi: 10.14740/gr913w. Epub 2017 Oct 26. PMID 29118867
- [Result] Gundermann KJ, Gundermann S, Drozdzik M, Mohan Prasad VG. Essential phospholipids in fatty liver: a scientific update. Clin Exp Gastroenterol. 2016 May 5;9:105-17. doi: 10.2147/CEG.S96362. eCollection 2016. PMID 27217791
- [Result] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183